CLINICAL TRIAL: NCT06561841
Title: A Multicenter, Randomized, Open-label Phase 2 Study to Evaluate the Efficacy and Safety of HSK39297 in Patients With Paroxysmal Nocturnal Hemoglobinuria（PNH）
Brief Title: A Study to Evaluate the Efficacy and Safety of HSK39297 in Patients With Paroxysmal Nocturnal Hemoglobinuria（PNH）
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSK39297-201
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2024-08

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental)
  Interventions: Drug: HSK39297
- Treatment group B (Experimental)
  Interventions: Drug: HSK39297
- Treatment group C (Experimental)
  Interventions: Drug: HSK39297

INTERVENTIONS:
Drug: HSK39297 — HSK39297 tablets for 24 weeks

SUMMARY:
This is a multicenter, randomized, open-label phase 2 study. Adult Patients with paroxysmal nocturnal hemoglobinuria naïve to complement inhibitor therapy were included. Subjects were treated with HSK39297 for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants ≥ 18 years of age;
2. Diagnosis of PNH based on flow cytometry with clone size > 10% by granulocytes;
3. Have not received complement inhibitor treatment;
4. Blood lactate dehydrogenase(LDH) values > 1.5 ×upper limit of the normal range (ULN) ;
5. Hemoglobin level < 100 g/L during the screening period.

Exclusion Criteria:

1. Hereditary or acquired complement deficiency;
2. Active primary or secondary immunodeficiency;
3. History of splenectomy, bone marrow/ hematopoietic stem cell or solid organ transplants;
4. History of recurrent invasive infections caused by encapsulated organisms( e.g. meningococcus or pneumococcus) or Mycobacterium tuberculosis;
5. Patients with laboratory evidence of bone marrow failure (reticulocytes < 100x10^9/L, or platelets < 30x10^9/L or neutrophils < 0.5x10^9/L) ;
6. Active systemic infection within 2 weeks prior to study drug administration;
7. History of serious comorbidities that have been determined to be unsuitable for participation in the study.
8. Pregnant or Lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with increase in hemoglobin levels from baseline of ≥20 g/L in the absence of red blood cell transfusions | Baseline, 24 weeks

SECONDARY OUTCOMES:
Proportion of participants with at least 60% reduction in LDH compared to baseline or LDH below the upper limit of normal | Baseline, 24 weeks
Change from baseline in hemoglobin | Baseline, 24 weeks
Change from baseline in reticulocyte count | Baseline, 24 weeks
Change from baseline in LDH | Baseline, 24 weeks
Change from baseline in Indirect bilirubin | Baseline, 24 weeks
Change from baseline in free hemoglobin | Baseline, 24 weeks
Proportion of participants without requiring red blood cells (RBC) transfusions | From week 4 to week 24
Change in the average number of RBC transfused per week | From week 4 to week 24
Change from baseline in PNH RBC clone size | Baseline, 24 weeks
Change from baseline in C3 fragment deposition on PNH RBC | Baseline, 24 weeks
Change from baseline in FACIT-Fatigue score | Baseline, 24 weeks
Incidence and severity of adverse events | 28 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No